CLINICAL TRIAL: NCT02741492
Title: Continuous Transversus Abdominus Plane Block for Open Inguinal Hernia Repair
Brief Title: Transversus Abdominus Plane Catheters for Open Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Neil Hanson, Staff Anesthesiologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Benaroya Research Institute
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Block Group (Active Comparator): Continuous Transversus Abdominis Plane Catheter
  Interventions: Procedure: Transversus Abdominis Plane Block
- Sham Group (Sham Comparator): Continuous Sham Catheter
  Interventions: Procedure: Sham Block

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — Continuous Nerve Block
  Arms: Block Group
Procedure: Sham Block — Continuous Sham Catheter
  Arms: Sham Group

SUMMARY:
This study is designed to evaluate pain control of continuous transversus abdominis plane (TAP) blocks placed for open inguinal hernia repair. The investigators hypothesize that there will be improved pain control when compared with sham blocks.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial designed to determine whether continuous transversus abdominis plane (TAP) block versus sham block has a substantial impact on pain following open inguinal hernia repair. Our primary outcome is to determine whether there will be a difference in opioid consumption within the first two days following surgery. Secondary outcomes will include: pain scores and activity assessment score.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral open inguinal hernia repair
* ASA physical status I-III
* >18 years old
* Consent to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* <18 years old
* Chronic opioid use
* Localized infection
* Pregnancy or lactating
* Pre-existing coagulopathy or active anticoagulant use
* Allergy to ultrasound gel or local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption (Intravenous Morphine Equivalents) | 48 Hours
  Total Opioid Consumption

SECONDARY OUTCOMES:
Pain (Numeric Rating) | 30 Days
  NRS Pain Scale
Activity Assessment Score | 30 Days
  Composite Score

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Hanson, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flaherty JM, Auyong DB, Yuan SC, Lin SE, Meier AW, Biehl TR, Helton WS, Slee A, Hanson NA. Continuous Transversus Abdominis Plane Block for Primary Open Inguinal Hernia Repair: A Randomized, Double-Blind, Placebo-Controlled Trial. Pain Med. 2020 Feb 1;21(2):e201-e207. doi: 10.1093/pm/pnz275. PMID 31670776